CLINICAL TRIAL: NCT00766129
Title: Comparison of Safety and Efficacy of Drug Eluting Stents : TAXUS (Boston Scientific) vs. LUC-Chopin (Balton, Poland) Implanted Into Saphenous Vein Grafts. Study With Serial Intravascular Ultrasounds.
Brief Title: Comparison of Safety and Efficacy of Two Different Drug Eluting Stents Implanted Into Saphenous Vein Grafts
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Adam Witkowski, Institute of Cardiology,Warsaw,Poland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N403 2786 33
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Stenosis in Saphenous Vein Graft, Drug Eluting Stent
Keywords: saphenous vein graft, TAXUS stent, Chopin stent

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- T (Experimental): Implantation of Taxus stent into saphenous vein graft
  Interventions: Device: Taxus stent implantation
- C (Experimental): Implantation of Luc-Chopin stent into saphenous vein graft
  Interventions: Device: Luc-Chopin stent

INTERVENTIONS:
Device: Taxus stent implantation — Patients will be treated with implantation of Taxus stent
  Arms: T
Device: Luc-Chopin stent — Patients will be treated will implantation of Luc-Chopin stent
  Arms: C

SUMMARY:
Drug eluting stents significantly reduced the rate of in-stent restenosis in coronary arteries. There are several kinds of DES i.e. eluting the drug either from stable or biodegradable polymer. The type of the polymer may impact the clinical outcome. The aim of our study was to compare safety and efficacy of implantation of two different types of stents eluting paclitaxel from stable vs biodegradable polymer (TAXUS stent vs LUC-CHOPIN stent) into coronary artery by-pass graft.

ELIGIBILITY:
Inclusion Criteria:

1. Atherosclerotic lesion in saphenous vein grafts causing angiographic stenosis ≥70%
2. Stable coronary artery disease or non ST segment elevation acute coronary syndrome
3. Reference segment diameter in range of 2.5-4.5mm

Exclusion Criteria:

1. Cardiogenic shock
2. Contraindications to prolonged dual antiplatelet therapy
3. Female of child birth potential unless on effective contraception
4. Other medical condition that may limit survival

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Neointima hyperplasia volume by Intravascular Ultrasound | 9 months

SECONDARY OUTCOMES:
All cause mortality | 5 years
Cardiovascular mortality | 5 years
Stent thrombosis | 5 years
Target lesion revascularization | 5 years
Angiographic late loss | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam R Witkowski, MD,PhD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, Warsaw, Poland